CLINICAL TRIAL: NCT00970905
Title: Effectiveness of Aprepitant in Addition to Ondansetron in the Prevention of Nausea and Vomiting Caused by Fractionated Radiotherapy to the Upper Abdomen
Brief Title: Effectiveness of Aprepitant in Addition to Ondansetron in the Prevention of Nausea and Vomiting Caused by Upper Abdominal Radiotherapy
Acronym: AVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Mayo Clinic (Other); Wake Forest University Health Sciences (Other); Norris Cotton Cancer Center (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Steven Ades, Assistant Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC 0908
Record Dates: First submitted 2009-08-25; First posted 2009-09-03 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Nausea; Vomiting
Keywords: Radiation; Nausea; Vomiting; Ondansetron; Aprepitant
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aprepitant & Ondansetron (Experimental)
  Interventions: Drug: aprepitant; Drug: Ondansetron

INTERVENTIONS:
Drug: aprepitant — aprepitant 125 mg po (Mondays), 80 mg po (Wednesdays), 80 mg po (Fridays) with doses scheduled 1-2 hours prior to the day's radiation fraction. Aprepitant will not be administered on weekend days. Aprepitant administration will continue until the last day of radiotherapy.
  Other Names: Emend
Drug: Ondansetron — Ondansetron 8 mg po bid, with the morning dose scheduled 1-2 hours prior to the day's radiation fraction. Ondansetron will not be administered on weekend days. Ondansetron administration will continue until the last day of radiotherapy.
  Other Names: Zofran

SUMMARY:
Severe nausea and/or vomiting in patients receiving radiotherapy to the upper abdomen is common despite having received pre-medication with ondansetron, a standard preventive treatment. This study aims to reduce the incidence of significant nausea and/or vomiting with the addition of the NK1-antagonist aprepitant to standard ondansetron treatment. This study will also assess the safety and tolerability of prolonged administration of aprepitant over the 4 to 6 week period of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a diagnosis of malignancy localized to the upper abdomen and requiring chemoradiation or radiation alone.
2. Receiving standard-fractionation radiation therapy (> 40 Gy) 3D-conformal radiation therapy or IMRT to a field involving the upper abdomen, either alone or combined with radiosensitizing 5FU, capecitabine, or gemcitabine permitted.
3. Age > 18 years old
4. Life expectancy >3 months
5. Performance status 0-2 inclusive
6. No more than mild to moderate hepatic impairment corresponding to Child-Pugh Class A or B, respectively (Child-Pugh score 5 to 9). See Appendix V for Child Pugh Classification.
7. Women of child-bearing potential and men must agree to use adequate contraception such as abstinence or effective barrier and/or non-hormonal contraception for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Adequate organ reserve to include: Absolute Neutrophil Count ≥ 1500/mcl , Hemoglobin ≥ 8.0 g/dl, platelet count ≥ 100,000/mcl, creatinine ≤ 2.0, AST & ALT ≤ 2.5 x ULN
9. Baseline ECG showing QTc value ≤ 480 millisecond
10. Informed consent

Exclusion Criteria:

1. Use of any other concomitant chemotherapy agent concurrently with radiation therapy aside from capecitabine, gemcitabine, or 5-fluorouracil (none of these agents are CYP 3A4 substrates).
2. Baseline vomiting is not controlled: Patients who have vomited or have nausea requiring antiemetic treatment within 24 hours prior to initiation of treatment.
3. Scheduled to receive treatment within 24 hours prior to day one or during the study periods with other potential or known antiemetic agents including but not limited to serotonin antagonists aside from ondansetron per study protocol, phenothiazines, butyrophenones, substituted benzamides, antihistamines, and cannabinoids. Chronically used benzodiazepines may be continued as a single nightly dose for sleep.
4. Any steroid use except topical steroids. Patients need to be off systemic steroid treatment for 7 days prior to start of chemoradiation therapy.
5. Uncontrolled CNS tumor
6. Other physical causes for nausea or vomiting (such as bowel obstruction) not related to chemoradiation administration
7. Hypersensitivity to either of the study agents
8. Planned simultaneous administration of any other investigational agents
9. Pregnant or nursing women
10. Patients taking other CYP3A4 inducers or inhibitors would be required to discontinue their use for at least 7 days prior to initiation of chemoradiation therapy. Examples of CYP3A4 inducers include aminoglutethimide, carbamazepine, nafcillin, nevirapine, phenobarbital, phenytoin, rifampin, and St. Johns Wort. Examples of CYP3A4 inhibitors include azole antifungals, clarithromycin, diclofenac, doxycycline, erythromycin, imatinib, isoniazid, nefazodone, nicardipine, propofol, protease inhibitors, quinidine, telithromycin, and verapamil.
11. CYP3A4 substrates are not contraindicated. However, patients taking CYP3A4 substrates should be cautioned to consult with their physician to minimize their use, if possible. Example substrates include benzodiazepines, calcium channel blockers, ranolazine, ergot derivatives, mirtazapine, nateglinide, tacrolimus, and venlafaxine.
12. Concomitant use of pimozide, terfenadine, cisapride, and astemizole is contraindicated per the Emend™ [10] product circular as dose-dependent inhibition of CYP 3A4 by aprepitant could result in elevated plasma concentrations of these drugs, potentially causing serious and life-threatening reactions. Patients taking these medications ineligible to participate in this study unless they are discontinued for at least 7 days prior to start of aprepitant.
13. Warfarin: Aprepitant may increase warfarin metabolism and the INR may be decreased. Twice weekly monitoring of INR recommended in the first 2-week period of radiation followed by weekly monitoring in subsequent weeks until discontinuation of aprepitant. Twice weekly monitoring is again recommended after aprepitant discontinuation until INR has stabilized.
14. Contraceptives (estrogens and progestins): Aprepitant may decrease the plasma levels of estrogen and progestin contraceptives. Contraceptive efficacy may be reduced. A nonhormonal form of contraception is necessary during treatment and for 1 month following the last dose of aprepitant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2016-07-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Complete Response rate (no vomiting and no rescue anti-emetic therapy) | overall period of radiation treatment (4-8 weeks)

SECONDARY OUTCOMES:
Complete Response rate | Cumulatively increasing time intervals from the start of radiation therapy (7 days, 14 days, 21 days, 28 days, 35 days, 42 days)
Proportion of patients who did not vomit | Overall period of radiation therapy (4-8 weeks)
No Significant Nausea: The proportion of patients who did not experience any nausea ≥ 3 on 0 - 10 scale | Overall period of radiation treatment (4-8 weeks)
No Nausea: The proportion of patients who did not experience any nausea. Nausea = 0 on 0 - 10 scale | Overall period of radiation treatment (4-8 weeks)
Complete Protection: The proportion of patients who did not vomit, require rescue therapy, or have nausea ≥ 3 on 0 - 10 scale | Overall period of radiation treatment (4-8 weeks)
Total Protection: The proportion of patients who did not vomit, require rescue therapy, or have any nausea (Nausea = 0 on 0 - 10 scale). | Overall period of radiation treatment (4-8 weeks)
Vomiting frequency: The frequency of vomiting (# episodes per week) in patients who did vomit at least once. | Overall period of radiation treatment (4-8 weeks)
Nausea frequency: The frequency of nausea (Nausea > 0 in a given week/ number of weeks during overall period of radiation treatment) | Overall period of radiation treatment (4-8 weeks)
Significant Nausea frequency: The frequency of significant nausea (Nausea ≥ 3 in a given week/ number of weeks during overall period of radiation treatment) | Overall period of radiation treatment (4-8 weeks)
Frequency of rescue medication use: The number of days in which rescue medication was taken / number of days of radiotherapy | overall period of radiation treatment (4-8 weeks)
Time to Failure: The time period in days from the start of radiation until the first vomiting episode or use of rescue medication for all patients and for the subset of patients who do not have a Complete Response. | Overall period of radiation treatment (4-8 weeks)
All adverse events that occur during radiation treatment with assessment of severity (CTC v.3) and relationship to study drug. | Overall period of radiation treatment (4-8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ades, MD MSc, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Derived] Ades S, Halyard M, Wilson K, Ashikaga T, Heimann R, Kumar S, Blackstock W. Effectiveness of aprepitant in addition to ondansetron in the prevention of nausea and vomiting caused by fractionated radiotherapy to the upper abdomen (AVERT). Support Care Cancer. 2017 May;25(5):1503-1510. doi: 10.1007/s00520-016-3540-4. Epub 2016 Dec 28. PMID 28032216